CLINICAL TRIAL: NCT03371979
Title: A Phase 1/2 Study of Pegzilarginase (AEB1102, Co-ArgI-PEG) in Combination With Pembrolizumab in the Treatment of Patients With Extensive Disease (ED) Small Cell Lung Cancer (SCLC)
Brief Title: Pegzilarginase and Pembrolizumab for Extensive Disease Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aeglea Biotherapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEB1102-101B; KEYNOTE PN758
Record Dates: First submitted 2017-11-20; First posted 2017-12-13 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegzilarginase plus Pembrolizumab (Experimental): Phase 1 & 2
  Interventions: Drug: Pegzilarginase; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pegzilarginase — Administered IV
  Other Names: AEB1102 (Co-ArgI-PEG)
Drug: Pembrolizumab — Administered IV
  Other Names: MK-3475; Keytruda

SUMMARY:
The main purpose of this Phase 1/2 study is to determine the safety and efficacy of pegzilarginase in combination with pembrolizumab in patients with ED-SCLC who have relapsed or progressive disease on or within 6 months of platinum-based chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient is able and willing to provide written informed consent
2. Be > 18 years of age on day of signing informed consent
3. Have histologically or cytologically confirmed SCLC that meets:

   1. Extensive disease per criteria of the International Association for the Study of Lung Cancer (IASLC)-American Joint Committee on Cancer (AJCC) TNM staging system
   2. Have not tolerated or have progressed or relapsed on or within 6 months of platinum-based chemotherapy
4. Have a performance status of ≤ 1 on the ECOG Performance Scale
5. Have measurable disease based on RECIST 1.1
6. Willing to undergo core needle or incisional biopsy to obtain fresh tumor tissue specimens
7. Demonstrate adequate organ function as evidenced by laboratory testing with specimens collected within 10 days prior to day 1 of cycle 1
8. Female child-bearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication
9. Sexually active male or female must be surgically sterile post-menopausal, or must agree to use a physician-approved method of birth control during the study through a minimum of 120 days after the last study drug administration.

Key Exclusion Criteria:

1. Has received more than 2 platinum-based regimens against SCLC
2. Has received pembrolizumab, or prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody as part of any previous therapy, including trials
3. Has participated in Merck MK-3475 (pembrolizumab) clinical trials
4. Has received pegzilarginase as part of any previous therapy
5. Is currently participating in a study of an investigational agent or received the last dose of an investigational agent within 4 weeks prior to the first dose of treatment in this study (a shorter interval for kinase inhibitors or other short half-life drugs could be considered after approval from the Sponsor). Is currently participating in a study of an investigational device within 4 weeks of the first dose of treatment
6. Has a diagnosis of an immunodeficiency, is receiving systemic steroid therapy (except for physiological dose levels), or immunosuppressive therapies
7. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer) that has undergone potentially curative therapy
8. Has known central nervous system (CNS) metastases. However, patients with previously treated brain metastases may participate provided neurologic symptoms have stabilized, there is no evidence of new brain metastases or hemorrhage and they are not using steroids for brain metastases or for complications derived from their treatment for at least 7 days prior to the first dose of trial treatment
9. Has known carcinomatous meningitis
10. Has an active autoimmune disease requiring systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs) or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections will not be excluded from the study. Patients with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment
11. Has evidence of interstitial lung disease, history of non-infectious pneumonitis that required steroids, or current pneumonitis
12. Inadequately controlled hypertension (defined as systolic blood pressure ≥ 200 mmHg and/or diastolic blood pressure ≥ 120 mmHg) on more than one occasion in the month before planned day of infusion
13. Currently taking 3 or more anti-hypertensive medications
14. Prior history of hypertensive crisis or hypertensive encephalopathy
15. History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or cardiac or vascular surgery within 6 months prior to day 1 of study treatment
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
17. Has a known history of Human Immunodeficiency Virus (HIV) (positive for HIV p24 antigen or HIV 1/2 antibodies)
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
19. Has a known history of active tuberculosis (Bacillus tuberculosis)
20. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
1. Phase 1: Incidence of treatment-related adverse events as assessed by CTCAE v4.0 | Estimated up to 6 months
  1. Number of participants experiencing treatment-related adverse events as assessed by CTCAE v4.0.
Phase 2: Efficacy determined by Objective Response Rate (ORR:CR+PR) per RECIST 1.1. | Estimated up to 6 months
  1. Objective Response Rate (ORR:) per RECIST 1.1
  • The Objective Response Rate (ORR) is defined as the percentage of subjects whose best objective response (BOR) is either complete response (CR) or partial response (PR). The ORR will be derived from the BOR according to response evaluation criteria in solid tumors (RECIST) v1.1 as assessed by the Investigator.

SECONDARY OUTCOMES:
Objective Response Rate | At 9, 18, and 27 weeks after first dose and every 12 weeks thereafter up to 24 months
  Percentage of patients whose cancer achieves either complete response (CR) or partial response (PR).
Clinical Benefit Rate | At 18 and 27 weeks after first dose and every 12 weeks thereafter up to 24 months
  Percentage of patients who have achieved CR, PR or Stable Disease (SD), lasting at least 8 weeks.
Time to Response | At 9, 18, and 27 weeks after first dose and every 12 weeks thereafter up to 24 months
  Time (weeks) from first treatment to the first documented CR or PR.
Duration of Response | At 18 and 27 weeks after first dose and every 12 weeks thereafter up to 24 months
  Time (weeks) from first documented CR or PR, until disease progression (PD).
Progression free survival | From first treatment up to 24 months
  Time (weeks) from first treatment to first observation of PD or death from any cause.
Overall Survival | From first treatment up to 24 months
  Time (weeks) from first treatment to death due to any cause.
Phase 2: Incidence of treatment-related adverse events as assessed by CTCAE v4.0 | From first treatment up to 24 months
  Number of participants experiencing treatment-related adverse events as assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Josie Gayton, Study Director — Aeglea Biotherapeutics, Inc.
Locations (22):
- United States (21):
  - University of Alabama, Mitchell Cancer Institute, Mobile, Alabama
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Mid Florida Hematology and Oncology Centers, Orange City, Florida
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - The Valley Hospital, Luckow Pavilion, Paramus, New Jersey
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - Providence Cancer Center, Portland, Oregon
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - West Clinic, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Memorial City, Houston, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Oncology & Hematology Associates of SW Virginia, Blacksburg, Virginia
- Fundacion De Investigacion, Hematology/Oncology, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No